CLINICAL TRIAL: NCT03443518
Title: Comparative Study Between Psoas Compartment Block (PCB) Versus Local Anesthesia With Remifentanil Infusion for Endovascular Repair of Abdominal Aortic Aneurysm (EVAR): A Randomized Controlled Trial
Brief Title: Psoas Compartment Block (PCB) Versus L.A Infiltration and Remifentanil Infusion During EVAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Erfan and Bagedo General Hospital (Other)
Responsible Party: Principal Investigator, DR. Osama Mohamed Farahat, Anesthesia consultant, Dr. Erfan and Bagedo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 180101
Record Dates: First submitted 2018-02-06; First posted 2018-02-23 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Analgesic Adverse Reaction
Keywords: EVAR, analgesia
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Local; Saline Solution; Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Physicians giving intraoperative care and recording data were blind to group type. Meanwhile, the anesthesiologist caring for the patient was aware to group type
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psoas Compartment Block (PCB) (Experimental): 30 ml of bupivacaine 0.25% will be infused over 3 minutes at the anatomical land mark for psoas plexus, also normal saline 0.9% IV infusion will be in the same rate of the Remifentanil infusion for the other group.
  Interventions: Procedure: Psoas Compartment Block (PCB); Drug: Normal saline 0.9% IV infusion
- L.A infiltration /Remifentanil infusion (Experimental): L.A infiltration (lidocaine) 5 ml of 2% will be injected subcutaneous as L.A infiltration then Remifentanil infusion with rate 0.03-0.1 μg / kg / min to achieve Visual Analog Scale 3 or less.
  Interventions: Procedure: Local Anesthesia infiltration; Drug: Remifentanil infusion

INTERVENTIONS:
Procedure: Psoas Compartment Block (PCB) — 30 ml of bupivacaine 0.25% will be infused over 3 minutes at the anatomical landmark for Psoas Compartment Block (PCB)
  Arms: Psoas Compartment Block (PCB)
Procedure: Local Anesthesia infiltration — Lidocaine 5 ml of 2% will be injected subcutaneous as local infiltration.
  Arms: L.A infiltration /Remifentanil infusion
Drug: Normal saline 0.9% IV infusion — Normal saline 0.9% IV infusion at the same rate of the Remifentanil infusion(0.05-0.1 μg/ kg/min).
  Arms: Psoas Compartment Block (PCB)
Drug: Remifentanil infusion — Remifentanil infusion with rate 0.03-0.1 μg/ kg/ min to achieve Visual Analog Scale (VAS) 3 or less
  Arms: L.A infiltration /Remifentanil infusion

SUMMARY:
Endovascular aneurysm repair (EVAR) was introduced in 1990 for the first time as a minimally invasive procedure instead of the conventional open surgical repair, with the aim to decrease morbidity and mortality . Nowadays EVAR has become an acceptable management for patients with infra-renal aortic aneurysms (AAA) . A lot of anesthetic techniques have been used successfully for EVAR. EVAR requires sedative analgesic medications to achieve an acceptable level of comfort to the patient and cardiorespiratory stability.

This is prospective randomized single blinded study of patients presenting with aorto-iliac aneurysm who will undergo EVAR. Patient's demographic data will be assessed, as well as clinical presentation, intraoperative complications.

30 patients undergoing elective EVAR will be included and will be divided equally into 2 groups.

First group is the psoas compartment block (PCB) (15 patients): 30 ml of bupivacaine 0.25% will be infused over 3 minutes at the anatomical landmark.

Second group is the LA and remifentanil group (LR) (15 patients): lidocaine 5 ml of 2% will be injected subcutaneous as local infiltration then remifentanil infusion with rate 0.03-0.1 μg kg-1 min-1. to achieve visual analog scale (VAS) 3 or less.

Vital date will be recorded as baseline then every 5 minutes till the end of the procedure. VAS will be recorded as baseline then every 5 minutes till the end of the procedure. Also stress response which will be measured subjectively as vital data and VAS and objectively as cortisol level in the blood which will be measured as base line and immediate after the end of the procedure.

DETAILED DESCRIPTION:
Anatomical, imaging and clinical studies suggest that psoas compartment block (PCB) which was done at L2-L3 level has a high possibility to include L1-L2 roots, and thus can be suitable for inguinal surgery. In our study, the investigators introduce a modified PCB which will be performed in lateral decubitus by a 120 mm stimulated needle inserted at the junction between the lateral third and the medial two-thirds of a line drawn at L2-L3 interspace, between the interspinous line and a line passing through the posterior superior iliac spine (PSIS), parallel to the interspinous line . If twitching of the anterior thigh area is observed, the needle is moved slight cranially. When twitching of the inguinal field is observed, bupivacaine 0.5% 30 ml, will be injected

ELIGIBILITY:
Inclusion Criteria:

* All elective patients presenting with aortoiliac aneurysm who will undergo percutaneous EVAR.

Exclusion Criteria:

* Exclusion criteria included the presence of an aneurysm of the common femoral artery or severe atherosclerotic disease with total occlusion, emergency EVAR, uncooperative patient, patient on anticoagulation therapy, cerebrovascular disease, poorly controlled hypertension (systolic arterial pressure ≥160 mmHg), poorly controlled diabetes mellitus (random blood glucose ≥200 mg/dL) and renal insufficiency (creatinine >1.5 mg/dL).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Changes in Visual Analogue Scale (VAS) | Assessment to be done at baseline (immediate before starting the procedure), then every 10 min through study till 4 hours after given the anesthesia.The event was determent via asking patient about pain experience every time using 100 mm VAS
  The primary outcome was Visual Analog Scale (VAS) to assess perioperative analgesia and pain management.
  Pain was assessed using the 100-mm visual analog scale, ranging from 0 to 100. The lowest score is 0 (no pain/excellent analgesia) and the highest score is 100 (Max pain).

SECONDARY OUTCOMES:
Arterial blood pressure | will be recorded at baseline (immediate before starting the procedure), then every 5 min through study till 4 hours after given the anesthesia.
  Arterial blood pressure monitoring in mmHg
Satisfactions Score | Time frame include 2 time points, first time point: immediate at the end of the procedure and the second time point: 2 hours after the end of the procedure
  Patient and surgeon satisfactions were assessed using the satisfaction score by asking them according to their degree of satisfaction based on this scale, which ranges from 0 to 100 (0 being the lowest score and 100 being the highest score).
heart rate (HR) | Will be recorded at baseline (immediate before starting the procedure), then every 5 min through study till 4 hours after given the anesthesia.
  heart rate monitoring in beat / min
Oxygen saturation | Will be recorded at baseline (immediate before starting the procedure), then every 5 min through study till 4 hours after given the anesthesia.
  Oxygen saturation monitoring in %

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - DR Erfan hospital, Jeddah
  - Erfan hospital, Jeddah

IPD SHARING:
Plan to Share IPD: Undecided